CLINICAL TRIAL: NCT04394923
Title: Impact of Pulmonary Vein Isolation (PVI) Line Modification Based on the Multidetector Computed Tomography (MDCT)-Derived Fingerprinted Esophageal Distance to the Posterior Wall of the Left Atrium, on the Esophageal Temperature Raise Measured With an Intraluminal Esophageal Temperature Monitoring Lead. A Randomized Controlled Study.
Brief Title: Relationship Between the Posterior Atrial Wall and the Esophagus: Esophageal Position and Temperature MEasurement During Atrial Fibrillation Ablation.
Acronym: AWESOME-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Head of the Arrhytmia Unit, Centro Medico Teknon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWESOME-AF
Record Dates: First submitted 2020-05-04; First posted 2020-05-20 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Atrial Arrhythmia
Keywords: Atrial fibrillation; Atypical flutter; catheter-based ablation; radiofrequency ablation; left atrial wall thickness; atrio-esophageal relationship
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Single center, prospective, randomized pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group or "PRINT" group (Experimental): The ablation line previously drawn will be modified regarding the esophageal print position in order to avoid RF application within the red layer of the esophageal print, which is the zone where the atrioesophageal distance is shorter. The maximal distance and the area between the original line and the modified line will be noted. In cases when ablation through the red layer is unavoidable, the delivered energy can be lowered to an ablation index (AI) of 300 regardless of the local wall thickness. If the temperature rises above 39℃, ablation will be immediately stopped, and energy will be reduced.
  Interventions: Procedure: Modification of the pulmonary vein ablation line
- Control group (Other): The ablation line will not be modified from the original one drawn before randomization and RF applications will follow the regular path. If the temperature rises above 39℃, ablation will be immediately stopped, and energy will be reduced.
  Interventions: Procedure: Regular PVI ablation

INTERVENTIONS:
Procedure: Modification of the pulmonary vein ablation line — The ablation line previously drawn will be modified regarding the esophageal print position in order to avoid RF application within the red layer of the esophageal print.
  Arms: Intervention group or "PRINT" group
Procedure: Regular PVI ablation — Blinded to the esophageal position based on the type of AF, closer to the ostium for paroxysmal AF and wider for persistent AF
  Arms: Control group

SUMMARY:
A multimodal strategy integrating esophageal visualization with the multidetector computed tomography (MDCT) and simultaneous temperature monitoring has never been put into practice. We have developed an isodistance map (esophageal print) to depict the atrio-esophageal relationship and to analyze the esophageal position peri procedurally. The present randomized study intends to analyze the usefulness of the esophageal print in predicting local thermal heating of the esophagus.

DETAILED DESCRIPTION:
Primary objective: to validate the usefulness of the esophageal print in avoiding temperature rises caused by radiofrequency (RF) application at the left atrial (LA) posterior wall during atrial fibrillation ablation

Secondary objectives:

1. to establish if there is a linear relationship between intraesophageal temperature rise and atrio-esophageal distance as calculated by the MDCT-derived esophageal print.
2. to analyze the need for ablation line modification.
3. to analyze the need for energy (power settings, ablation index, ablation time, etc.) modification.
4. to develop a new multimodal approach to esophageal monitoring during AF/AT ablation.

Interventions

1. Pre-procedural scan and Esophageal Isodistance Print

   The methods for the acquisition of the cardiac MDCT and the image processing have been described in Part 1. During the segmentation process, the epicardial layer of the posterior atrial wall and the esophageal wall have been defined. The distance between these two structures is computed at each epicardial point, allowing to create an esophageal print on top of the epicardial layer. The isodistance color map uses a color scale to depict a range of distance; red being the closest (< 1 mm) and purple being the most distant (> 4 mm). Yellow, green and blue will be considered the intermediate values.
2. Luminal esophageal temperature (LET) monitoring

   A multi-thermocouple temperature probe (SensiTherm, St. Jude Medical, Inc., St. Paul, MN, USA) will be advanced via transnasal or transoral access into the esophagus once the patient is under general anesthesia. When the esophageal print is close to the ablation line, the temperature probe position will be adjusted under fluoroscopic guidance before application at each pair of pulmonary veins to ensure that it overlaps the ablation line. All esophageal temperature rises above 39 °C will be documented and RF application will be stopped.
3. Pulmonary vein ablation lines regarding Esophageal Isodistance Print

Before randomization, an investigator blinded to the esophageal position will draw the PVI ablation line around both pairs of veins based on the type of AF (closer to the ostium for paroxysmal AF and wider for persistent AF).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Indication for any atrial fibrillation or left atrial flutter ablation procedure.
* Documented episodes of atrial arrhythmia (AF/AT/AFL)
* Signed informed consent.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Impossibility to perform CT Scan.
* Impossibility to perform transesophageal echocardiography or to insert esophageal temperature monitoring probe.
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical
* Inability to give written informed consent.
* Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants presenting a temperature rise as measured with a luminal esophageal temperature probe during radiofrequency delivery. The temperature is measured in Celsius degrees. | 1 day
  Number of intraesophageal temperature rises above 39°C or absolute temperature raises of 2°C degrees. The chosen probe is St Jude

SECONDARY OUTCOMES:
Proportion of patients needing ablation power or ablation time modification owing to esophageal presence in the immediate posterior wall . | 1 day
  Modification of the ablation parameters.Power is measured in Watts during radiofrequency application. Ablation time is measured in seconds of radiofrequency application. Both measures are provided by the electroanatomical navigation system.

CONTACTS AND LOCATIONS:
Locations (1):
- Teknon Medical Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Suenari K, Nakano Y, Hirai Y, Ogi H, Oda N, Makita Y, Ueda S, Kajihara K, Tokuyama T, Motoda C, Fujiwara M, Chayama K, Kihara Y. Left atrial thickness under the catheter ablation lines in patients with paroxysmal atrial fibrillation: insights from 64-slice multidetector computed tomography. Heart Vessels. 2013 May;28(3):360-8. doi: 10.1007/s00380-012-0253-6. Epub 2012 Apr 22. PMID 22526381
- [Background] Sanchez-Quintana D, Cabrera JA, Climent V, Farre J, Mendonca MC, Ho SY. Anatomic relations between the esophagus and left atrium and relevance for ablation of atrial fibrillation. Circulation. 2005 Sep 6;112(10):1400-5. doi: 10.1161/CIRCULATIONAHA.105.551291. Epub 2005 Aug 29. PMID 16129790
- [Background] Lakkireddy D, Reddy YM, Atkins D, Rajasingh J, Kanmanthareddy A, Olyaee M, Dusing R, Pimentel R, Bommana S, Dawn B. Effect of atrial fibrillation ablation on gastric motility: the atrial fibrillation gut study. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):531-6. doi: 10.1161/CIRCEP.114.002508. Epub 2015 Mar 14. PMID 25772541
- [Background] Lemola K, Sneider M, Desjardins B, Case I, Han J, Good E, Tamirisa K, Tsemo A, Chugh A, Bogun F, Pelosi F Jr, Kazerooni E, Morady F, Oral H. Computed tomographic analysis of the anatomy of the left atrium and the esophagus: implications for left atrial catheter ablation. Circulation. 2004 Dec 14;110(24):3655-60. doi: 10.1161/01.CIR.0000149714.31471.FD. Epub 2004 Nov 29. PMID 15569839
- [Background] Tsao HM, Wu MH, Higa S, Lee KT, Tai CT, Hsu NW, Chang CY, Chen SA. Anatomic relationship of the esophagus and left atrium: implication for catheter ablation of atrial fibrillation. Chest. 2005 Oct;128(4):2581-7. doi: 10.1378/chest.128.4.2581. PMID 16236927
- [Background] Kennedy R, Good E, Oral H, Huether E, Bogun F, Pelosi F, Morady F, Chugh A. Temporal stability of the location of the esophagus in patients undergoing a repeat left atrial ablation procedure for atrial fibrillation or flutter. J Cardiovasc Electrophysiol. 2008 Apr;19(4):351-5. doi: 10.1111/j.1540-8167.2007.01051.x. Epub 2007 Dec 12. PMID 18081769
- [Background] Starek Z, Lehar F, Jez J, Scurek M, Wolf J, Kulik T, Zbankova A. Esophageal positions relative to the left atrium; data from 293 patients before catheter ablation of atrial fibrillation. Indian Heart J. 2018 Jan-Feb;70(1):37-44. doi: 10.1016/j.ihj.2017.06.013. Epub 2017 Jun 29. PMID 29455785
- [Background] Barbhaiya CR, Kumar S, Guo Y, Zhong J, John RM, Tedrow UB, Koplan BA, Epstein LM, Stevenson WG, Michaud GF. Global Survey of Esophageal Injury in Atrial Fibrillation Ablation: Characteristics and Outcomes of Esophageal Perforation and Fistula. JACC Clin Electrophysiol. 2016 Apr;2(2):143-150. doi: 10.1016/j.jacep.2015.10.013. Epub 2015 Dec 23. PMID 29766863
- [Background] Halbfass P, Pavlov B, Muller P, Nentwich K, Sonne K, Barth S, Hamm K, Fochler F, Mugge A, Lusebrink U, Kuhn R, Deneke T. Progression From Esophageal Thermal Asymptomatic Lesion to Perforation Complicating Atrial Fibrillation Ablation: A Single-Center Registry. Circ Arrhythm Electrophysiol. 2017 Aug;10(8):e005233. doi: 10.1161/CIRCEP.117.005233. PMID 28798021
- [Background] Kapur S, Barbhaiya C, Deneke T, Michaud GF. Esophageal Injury and Atrioesophageal Fistula Caused by Ablation for Atrial Fibrillation. Circulation. 2017 Sep 26;136(13):1247-1255. doi: 10.1161/CIRCULATIONAHA.117.025827. PMID 28947480
- [Background] Zellerhoff S, Ullerich H, Lenze F, Meister T, Wasmer K, Monnig G, Kobe J, Milberg P, Bittner A, Domschke W, Breithardt G, Eckardt L. Damage to the esophagus after atrial fibrillation ablation: Just the tip of the iceberg? High prevalence of mediastinal changes diagnosed by endosonography. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):155-9. doi: 10.1161/CIRCEP.109.915918. Epub 2010 Mar 1. PMID 20194799
- [Background] Kadado AJ, Akar JG, Hummel JP. Luminal esophageal temperature monitoring to reduce esophageal thermal injury during catheter ablation for atrial fibrillation: A review. Trends Cardiovasc Med. 2019 Jul;29(5):264-271. doi: 10.1016/j.tcm.2018.09.010. Epub 2018 Sep 19. PMID 30282588
- [Background] Kaneshiro T, Matsumoto Y, Nodera M, Kamioka M, Kamiyama Y, Yoshihisa A, Ohkawara H, Suzuki H, Takeishi Y. Anatomical predisposing factors of transmural thermal injury after pulmonary vein isolation. Europace. 2018 Jul 1;20(7):1122-1128. doi: 10.1093/europace/eux185. PMID 28605437
- [Background] Kottkamp H, Piorkowski C, Tanner H, Kobza R, Dorszewski A, Schirdewahn P, Gerds-Li JH, Hindricks G. Topographic variability of the esophageal left atrial relation influencing ablation lines in patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2005 Feb;16(2):146-50. doi: 10.1046/j.1540-8167.2005.40604.x. PMID 15720452
- [Derived] Teres C, Soto-Iglesias D, Penela D, Falasconi G, Viveros D, Meca-Santamaria J, Bellido A, Alderete J, Chauca A, Ordonez A, Marti-Almor J, Scherer C, Panaro A, Carballo J, Camara O, Ortiz-Perez JT, Berruezo A. Relationship between the posterior atrial wall and the esophagus: esophageal position and temperature measurement during atrial fibrillation ablation (AWESOME-AF). A randomized controlled trial. J Interv Card Electrophysiol. 2022 Dec;65(3):651-661. doi: 10.1007/s10840-022-01302-0. Epub 2022 Jul 21. PMID 35861901